CLINICAL TRIAL: NCT03689920
Title: Study to Demonstrate the Value of Multiple Modalities and Combining Mechanisms Using the Spectra WaveWriter™ Spinal Cord Stimulator System in the Treatment of Chronic Pain
Brief Title: Combining Mechanisms for Better Outcomes (COMBO)
Acronym: COMBO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A4070
Record Dates: First submitted 2018-09-27; First posted 2018-10-01 (Actual); Results first posted 2020-11-27 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Chronic Pain; Back Pain
MeSH Terms: conditions — Chronic Pain; Back Pain | interventions — Spinal Cord Stimulation; Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- WaveWriter Settings (Active Comparator): WaveWriter Programming
  Interventions: Device: Boston Scientific Spectra WaveWriter™ Spinal Cord Stimulation (SCS) System
- Conventional Settings (Active Comparator): Conventional Programming
  Interventions: Device: Boston Scientific Spectra WaveWriter™ Spinal Cord Stimulation (SCS) System

INTERVENTIONS:
Device: Boston Scientific Spectra WaveWriter™ Spinal Cord Stimulation (SCS) System — The Spectra WaveWriter Spinal Cord Stimulator (SCS) System is indicated as an aid in the management of chronic intractable pain of the trunk and/or limbs, including unilateral or bilateral pain associated with the following: failed back surgery syndrome, Complex Regional Pain Syndrome (CRPS) Types I and II, intractable low back pain and leg pain.

SUMMARY:
To evaluate the effectiveness of Spinal Cord Stimulation (SCS) with multiple modalities as compared to conventional SCS in patients with chronic pain when using the Boston Scientific Spectra WaveWriter SCS System.

DETAILED DESCRIPTION:
To evaluate the effectiveness of Spinal Cord Stimulation (SCS) with multiple modalities as compared to conventional SCS in patients with chronic pain when using the Boston Scientific Spectra WaveWriter SCS System.

ELIGIBILITY:
Key Inclusion Criteria:

* Chronic pain of the trunk and/or limbs for at least 6 months with back pain greater or equal to leg pain.
* 22 years of age or older at time of enrollment
* Able to independently read and complete all questionnaires and assessments provided in English
* Signed a valid, IRB-approved informed consent form (ICF) provided in English

Key Exclusion Criteria:

* Any pain-related diagnosis or medical/psychological condition that, in the clinician's best judgment, might confound reporting of study outcomes
* Significant cognitive impairment that, in the opinion of the Investigator, would reasonably be expected to impair the study candidate's ability to participate in the study
* Breast-feeding or planning to get pregnant during the course of the study or not using adequate contraception
* Participating, or intends to participate, in another clinical trial that may influence the data that will be collected for this study

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2018-10-03 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2021-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Wallace, M.D., Principal Investigator — University of California, San Diego
Locations (15):
- United States (15):
  - Center for Pain and Supportive Care, Phoenix, Arizona
  - UCSD Medical Center - Jacobs Medical Center, La Jolla, California
  - Denver Back Pain Specialists, Greenwood Village, Colorado
  - South Lake Pain Institute, Inc, Clermont, Florida
  - Willis-Knighton River Cities Clinical Research Center, Shreveport, Louisiana
  - Michigan Pain Consultants, Grand Rapids, Michigan
  - Forest Health Medical Center, Ypsilanti, Michigan
  - KC Pain Centers, Lee's Summit, Missouri
  - Carolinas Research Institute, LLC, Huntersville, North Carolina
  - The Center for Clinical Research, LLC, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Toledo Clinic, Toledo, Ohio
  - Pacific Sports and Spine, LLC, Eugene, Oregon
  - Precision Spine Care, Tyler, Texas
  - EvergreenHealth Pain Care, Kirkland, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wallace MS, North JM, Phillips GM, Calodney AK, Scowcroft JA, Popat-Lewis BU, Lee JM, Washabaugh EP 3rd, Paez J, Bolash RB, Noles J, Atallah J, Shah B, Ahadian FM, Trainor DM, Chen L, Jain R. Combination therapy with simultaneous delivery of spinal cord stimulation modalities: COMBO randomized controlled trial. Pain Manag. 2023 Mar;13(3):171-184. doi: 10.2217/pmt-2022-0101. Epub 2023 Mar 3. PMID 36866658

RESULTS

PARTICIPANT FLOW:
Recruitment Details: After subjects were enrolled, they were evaluated per study eligibility criteria. Only those who met all criteria proceeded to receive implant and randomized in the study (as applicable).
Period: Overall Study
Arm/Group | WaveWriter Settings | Conventional Settings
Started | 47 | 52
Completed | 41 | 48
Not Completed | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | WaveWriter Settings | Conventional Settings | Total
Number analyzed (Participants) | 47 | 52 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (12.23) | 57.8 (12.09) | 57.1 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 36 | 66
  Male | 17 | 16 | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black, of African Heritage | 0 | 1 | 1
  Caucasian | 47 | 49 | 96
  Hispanic or Latino | 0 | 1 | 1
  Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Pain Responder Rate
Description: Percentage of subjects with 50% or greater reduction from Baseline Visit in average overall pain intensity at 3 months post-randomization with no increase in opioid medications
Time Frame: 3 months post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | WaveWriter Settings | Conventional Settings
Number analyzed (Participants) | 41 | 48
Participants | 36 | 34

ADVERSE EVENTS:
Time Frame: Adverse Events were collected up to end of randomized phase (3 months post-randomization)
Description: Adverse Events including Serious Adverse Events were collected up to end of randomized phase (3 months post-randomization)
Arm/Group | WaveWriter Settings | Conventional Settings
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/48
Serious Adverse Events (participants affected / at risk) | 4/41 | 5/48
Other Adverse Events (participants affected / at risk) | 0/41 | 0/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | WaveWriter Settings (N=41) | Conventional Settings (N=48)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Carotid Artery Stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic Stroke (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-31): https://cdn.clinicaltrials.gov/large-docs/20/NCT03689920/Prot_SAP_000.pdf